CLINICAL TRIAL: NCT02865356
Title: Evaluation of SP14019-F-01 Topical Solution for the Treatment of Atopic Dermatitis. Pilot Study (CYCLATOP STUDY)
Brief Title: Topical Solution for the Treatment of Atopic Dermatitis
Acronym: CYCLATOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spherium Biomed (Industry)
Collaborators: Germans Trias i Pujol Hospital (Other); Hospital del Mar (Other); Hospital Sant Joan de Deu (Other); Hospital Universitario Virgen Macarena (Other); Hospital Universitario La Fe (Other); Hospital General Universitario de Alicante (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Hospital Universitario Virgen de la Victoria (Other); Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP14019-18
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; eczema; children; skin; topical; cyclosporine
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Cyclosporine; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclosporine 5% Solution (Experimental): SP14019-F-01 Cyclosporine solution, 5%. Cyclosporine solution will be applied twice daily for four complete weeks (28 days) in all affected areas.
  A randomized list will be created to determine in which side of the body (left or right) the subject will apply each medication
  Interventions: Drug: Cyclosporine 5% solution
- Placebo (Placebo Comparator): SP14019-F-02 vehicle-control placebo solution. Vehicle-control placebo solution will be applied twice daily for four complete weeks (28 days) in all affected areas.
  A randomized list will be created to determine in which side of the body (left or right) the subject will apply each medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyclosporine 5% solution — topical solution
  Other Names: ciclosporin
  Arms: Cyclosporine 5% Solution
Drug: Placebo — topical vehicle solution
  Other Names: SP14019-F-02 Placebo
  Arms: Placebo

SUMMARY:
The study is designed as a proof of concept, multi-center, randomized, double-blind and vehicle-controlled study with intra-individual comparison of treatments.

Three age cohorts of patients will be included in the study according to the following age ranges:

1. ≥18 years old (minimum 6, maximum 18 patients)
2. >12 - 17 years old (minimum 6, maximum 18 patients)
3. >2 - 12 years old (minimum 6, maximum 18 patients)

The main objectives of study are:

To assess the efficacy of SP14019-F-01 topical solution (5% cyclosporine A [CsA]) compared to placebo topical solution for the treatment of patients with mild to moderate atopic dermatitis (AD).

To evaluate the safety and tolerability of SP14019-F-01 (5% CsA) topical solution in patients with mild to moderate AD.

DETAILED DESCRIPTION:
The study is designed as a proof of concept, multi-center, randomized, double-blind and vehicle-controlled study with intra-individual comparison of treatments. CsA plasma concentration assessments will be carried out at Visit 0 predose, and Visits 1 and 4 of the study period.

Three age cohorts of patients will be included in the study according to the following age ranges:

1. ≥18 years old (minimum 6, maximum 18 patients)
2. >12 - 17 years old (minimum 6, maximum 18 patients)
3. >2 - 12 years old (minimum 6, maximum 18 patients) The study will close when the total of 36 patients has been included among all age groups and the minimum number of 6 patients has been reached for each age group.

Before including paediatric population, a minimum of 6 adult patients should complete the treatment to assess the safety profile.

A randomized list will be created to determine in which side of the body (left or right) the subject will apply each medication (SP14019-F-01 topical solution [5% CsA] or SP14019-F-02 vehicle-control placebo solution). Solutions will be applied twice daily for four complete weeks (28 days) in all affected areas.

Photography will be used to record the evolution of the lesions at Visits 0 (pre-1st dose), Visits 1, 2, 3, 4 and follow-up.

The main objectives of study are:

To assess the efficacy of SP14019-F-01 topical solution (5% cyclosporine A [CsA]) compared to placebo topical solution for the treatment of patients with mild to moderate atopic dermatitis (AD).

To evaluate the safety and tolerability of SP14019-F-01 (5% CsA) topical solution in patients with mild to moderate AD.

A Steering Committee will convene periodically to maintain the quality of study conduct, and to discuss any major issues or concerns and with particular attention to some critical events which may lead to stop the recruitment. These critical events are the observation of either new unexpected signals on safety related to CsA. The Steering Committee will also evaluate the safety profile of the treatment before including paediatric population

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 2 and 75 years, inclusive, at the screening visit. 2. AD diagnosis according to the Hanifin/Rajka criteria with one eczema outbreak at the screening and baseline.

  3. Presence of at least two lesional areas. These areas should be at the left and right side of the body and occupying a body surface area (BSA) in each side between 0.1% and 10% of the BSA. IGA score of the two sites not differ by more than 1 point.

  4. Mild to moderate disease severity of AD defined by an IGA score of 2 or 3 at baseline (IGA scale from 0 to 4).

  5. Total BSA of AD involvement ≤ 10% in each side of the body (≤ 20% maximum). 6. Normal weight as defined by a Quetelet Index (Body Mass Index [BMI]: weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2 (both included).

  7. General medical condition, in the investigator's opinion, does not interfere with the assessments and the completion of the trial.

  8. Parent's or legal guardian's written informed consent and child assent, if appropriate or patient's inform consent for patients ≥ 18 years of age before any assessment is performed.

  9. Able to communicate with the investigator and comply with the requirements of the study (for children the parent can assist when necessary).

Exclusion Criteria:

* 1. Female subject of childbearing potential without use of effective birth control methods, or not willing to continue practicing these birth control methods for at least 30 days after the end of the treatment period;

Note: Estrogen based hormonal contraception may not be reliable when SP14019-F-01 topical solution is applied, therefore to be eligible for this trial, women of childbearing potential should either:

1. use a double barrier method to prevent pregnancy (i.e., using a condom with either diaphragm or cervical cap);
2. use hormonal based contraceptives in combination with a barrier contraceptive (i.e., male condom, diaphragm or cervical cap, or female condom);
3. use an intrauterine device in combination with a barrier contraceptive (i.e., male condom, diaphragm or cervical cap, or female condom);
4. be only non-heterosexually active, practice heterosexual abstinence, or have a vasectomized partner (confirmed sterile). Women with tubal ligation are required to use 1 non-hormonal contraceptive method.

   Women who are postmenopausal for at least 2 years, and women with total hysterectomy are considered of non-childbearing potential. Males with partners of childbearing potential should inform them of their participation in this clinical study and use a highly effective method of birth control during the study.

   2. Pregnant woman or with a positive pregnancy test or breast feeding at baseline.

   3. Any condition in the lesions that in the opinion of the investigator could interfere with clinical assessments, e.g. acne, infection, rash other than AD, sunburn, scars, hairy or tattooed area.

   4. Patients receiving phototherapy or systemic therapy for AD within 4 weeks before the first application of trial medication.

   5. Patients receiving antibiotics, topical therapy for AD within 2 weeks before the first application of trial medication.

   6. Patients taking antihistamines within 1 week before the first application of trial medication.

   7. Patients receiving radiation therapy, systemic therapy with cytostatics or biological therapy within 24 weeks before the first application of trial medication, or with previous history of malignancy (excluding basal cell carcinoma).

   8. Patients with any acute skin infection (superinfection or secondary impetiginisation).

   9. Patients with confirmed hypertension, renal disease or serious infections at screening.

   10. Any currently active allergy such as but not limited to drug allergy, food allergy or hay fever.

   11. Previously demonstrated clinically significant allergy or hypersensitivity to any of the excipients of the trial medication administered in this trial.

   12. Participation in an investigational drug trial within 30 days prior to the first application of trial medication.

   13. Any condition (including but not limited to alcohol and drug use), which in the opinion of the investigator could compromise the patient safety or compliance with trial procedures.

   14. Subjects who have received or are planning to receive any vaccination within 28 days prior to the first dose of study medication, or planning to receive a vaccination during the course of the study.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline (Day 0) of Eczema Area and Severity Index (EASI) score of the treated body area (CsA vs Vehicle control placebo) | Absolute change from Day 0 (baseline) to Day 7 (Visit 1), Day 14 (Visit 2), Day 21(Visit 3) and Day 28 (Visit 4).
Change from baseline (Day 0) of Investigator's Global Assessment (IGA) score (on a 0 to 4-point scale; CsA vs Vehicle control placebo) | Absolute change from Day 0 (baseline) to Day 7 (Visit 1), Day 14 (Visit 2), Day 21(Visit 3) and Day 28 (Visit 4).
Absolute change from baseline (Day 0) of Atopic Dermatitis Severity Index (ADSI) score (Cs vs Vehicle control placebo) | Absolute change from Day 0 (baseline) to Day 7 (Visit 1), Day 14 (Visit 2), Day 21(Visit 3) and Day 28 (Visit 4).

SECONDARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events (TEAEs). | From date of randomization (Day 0) until 6 weeks
Frequency and severity of TEAEs leading to study drug discontinuation | From date of randomization (Day 0) until 6 weeks
CsA plasma concentrations | From date of randomization (Day 0) up to 4 weeks, on day 7 and 28.
  samples obtained just before the first daily dose (around 8 am) on Visits 0, 1 and 4 to check the absence of systemic absorption during the period of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ferrándiz, MD, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (9):
- Spain (9):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided